CLINICAL TRIAL: NCT00531674
Title: Efficacy of 3 Nutritional Supplements to Improve Diverse Outcomes in Children Under 2 Years of Age and Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mexican National Institute of Public Health (Other Government)
Collaborators: Secretary of Social Development (Unknown); Inter-American Development Bank (Other)
Responsible Party: Armando Garcia Guerra, National Institute of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NIPH472
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Efficacy of public health intervention (nutrition)
MeSH Terms: interventions — Gravidity; Tablets

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nutritional supplementation for pregnant and lactating women
  Interventions: Dietary Supplement: fortified milk-based beverage; Dietary Supplement: Sprinkles; Dietary Supplement: tablets
- 2 (Experimental): Nutritional supplementation for children
  Interventions: Dietary Supplement: Fortified milk-based pap; Dietary Supplement: Sprinkles; Dietary Supplement: Syrup

INTERVENTIONS:
Dietary Supplement: fortified milk-based beverage — Fortified with multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for women.
  Other Names: Nutrivida
  Arms: 1
Dietary Supplement: Sprinkles — Powder with multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for women.
  Other Names: Vita-mine for pregnant and lactating women
  Arms: 1
Dietary Supplement: tablets — Multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for women.
  Arms: 1
Dietary Supplement: Fortified milk-based pap — Fortified with multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for children.
  Other Names: Nutrisano
  Arms: 2
Dietary Supplement: Sprinkles — Powder with multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for women.
  Other Names: Vita-mine for children
  Arms: 2
Dietary Supplement: Syrup — Multiple vitamins and minerals (1 RDA). Identifical dose and formulation as other supplements for women.
  Arms: 2

SUMMARY:
The Mexican poverty alleviation program, Oportunidades provides a fortified food supplement to all beneficiary children under 2 years of age, and all pregnant and lactating women. Consumption of the supplements is well below recommended levels and the impact of the program on child growth and anemia is less than anticipated. This is likely due to a high degree of dilution by sharing of the supplements with other family members. We have also found evidence of a very high prevalence of overweight and obesity among beneficiaries of Oportunidades in both women and children.

Given the micronutrient content of the fortified food, it is likely that the impact of the program on child growth and the micronutrient status of women and children would improve considerable if the supplements were consumed daily in the recommended dose. This may be difficult, given the wide-spread sharing within households - something that has been identified by many beneficiary families as a desirable behavior. At the same time, we do not know whether daily consumption of the food, which contains approximately 20% of daily energy requirements, may contribute to undesirable weight gain in this population.

In this context, we have designed a cluster randomized controlled efficacy trail to compare the nutritional impact, acceptability and use of three nutritional supplements. Supplements were randomly assigned at the community level (n=54), and pregnant women (n=750) and children 6 to 12 mo of age (n=900) invited to participate. The principal objective of the study is to compare the impact of Sprinkles and Nutrisano/Nutrivida using syrup/pills as a positive control group, on child growth, weight gain and retention in pregnant women, and micronutrient status of women and children. We hypothesize that weight gain will be greater in the food group compared to the other two supplementation groups, but impacts on micronutrient status and length growth in children will be similar.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women before 27 wks pregnancy (Arm 1)
* 18 yrs of age and older (Arm 1)
* Children 6 to 12 mo of age (Arm 2)
* Beneficiaries of the Oportunidades programa (Arm 1 and 2)

Exclusion Criteria:

* Severe anemia (Arm 1 and 2)
* Consuming other nutritional supplements and unwilling to descontinue use (Arm 1 and 2)

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Child linear growth and weight gain | 24 mo of age
  Child height and weight at 24 mo of age and increment from baseline to 24 mo of age
Child hemoglobin concentration and anemia prevalence | 10 mo of supplementation, at 24 mo of age, 6 mo after completion of supplementation (30 mo of age)
Pregnancy weight gain and weight retention | 37 wks pregnancy, 1 and 3 mo postpartum
Hemoglobin concentration and anemia prevalence | 37 wks pregnancy and 1 mo postpartum

SECONDARY OUTCOMES:
Acceptability and use of the supplements (women and children) | Children: after 2, 6 and 12 mo consumption; Women: following completion of trial and in pregnant women who did not participate in main study
Physical activity in children | after 4 and 12 mo of supplementation
Language adquisition and motor milestone development in children | Throughout follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette M Neufeld, PhD, Principal Investigator — National Institute of public Health

REFERENCES:
- [Derived] Neufeld LM, Garcia-Guerra A, Quezada AD, Theodore F, Bonvecchio Arenas A, Islas CD, Garcia-Feregrino R, Hernandez A, Colchero A, Habicht JP. A Fortified Food Can Be Replaced by Micronutrient Supplements for Distribution in a Mexican Social Protection Program Based on Results of a Cluster-Randomized Trial and Costing Analysis. J Nutr. 2019 Dec 1;149(Suppl 1):2302S-2309S. doi: 10.1093/jn/nxz176. PMID 31793645
- See also: Home page, National Institute of Public Health, Mexico — http://www.insp.mx